CLINICAL TRIAL: NCT04752436
Title: Supra High-intensity Interval Training for Austin Police Officers
Brief Title: Supra High-intensity Interval Training for Police Officers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019090050
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Physical Fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supra high intensity interval training (Experimental): The experimental group will engage in the high intensity interval training.
  Interventions: Behavioral: Supra high intensity interval training

INTERVENTIONS:
Behavioral: Supra high intensity interval training — The exercise program will consist of eight 20-second all-out exercise bouts followed by 10 seconds of rest for a total of 4 minutes of total exercise duration. The intensity of exercise is all out. The exercise will be conducted 3 times a week for 8 weeks.

SUMMARY:
Police work is extreme in terms of the physical activity and physical exertion spectrum as it is composed of a mixture of enforced sitting and sudden physical exertion. Police officers remain sitting for the majority of their working hours. In theory, regular physical activity exerts a number of health and fitness benefits that could act on most issues that police officers suffer from. Supra high-intensity interval training (supra HIIT) appears to be a perfect solution for police officers as the training modality can be accomplished in less than 5 minutes. The primary purpose of this proposal is to create and assess supra HIIT program that is suitable for police officers and then to assess feasibility of such exercise program in a small pilot study.

ELIGIBILITY:
Inclusion Criteria:

• Police officers in the local Police Department who are capable of performing physical exercise

Exclusion Criteria:

* Being pregnant
* Having had a recent illness
* History of diabetes, heart disease, or other cardiovascular problems
* Recent surgery, orthopedic, or musculoskeletal injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Aerobic power | 8 weeks
  Aerobic fitness or maximal oxygen consumption will be evaluated during incremental treadmill exercise tests (1% grade increase per minute at individualized treadmill speed).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Masked data will be shared by other investigators with a reasonable request following the publication of the data.